CLINICAL TRIAL: NCT00003643
Title: Randomized Phase II/III Study of Taxol/Paclitaxel-BEP Versus BEP in Patients With Intermediate Prognosis Germ Cell Cancer
Brief Title: Combination Chemotherapy in Treating Men With Germ Cell Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-30983; EORTC-30983
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-03

CONDITIONS: Extragonadal Germ Cell Tumor; Teratoma; Testicular Germ Cell Tumor
Keywords: stage III malignant testicular germ cell tumor; testicular seminoma; testicular embryonal carcinoma; testicular choriocarcinoma; testicular yolk sac tumor; testicular embryonal carcinoma and teratoma; testicular embryonal carcinoma and teratoma with seminoma; testicular embryonal carcinoma and yolk sac tumor; testicular embryonal carcinoma and yolk sac tumor with seminoma; testicular embryonal carcinoma and seminoma; testicular yolk sac tumor and teratoma; testicular yolk sac tumor and teratoma with seminoma; testicular choriocarcinoma and yolk sac tumor; testicular choriocarcinoma and embryonal carcinoma; testicular choriocarcinoma and teratoma; testicular choriocarcinoma and seminoma; stage IV extragonadal non-seminomatous germ cell tumor; stage IV extragonadal seminoma; testicular immature teratoma; testicular mature teratoma; adult teratoma
MeSH Terms: conditions — Teratoma; Testicular Germ Cell Tumor; Testicular Neoplasms; Seminoma; Endodermal Sinus Tumor; Carcinoma, Embryonal | interventions — Bleomycin; Filgrastim; Cisplatin; Etoposide; Paclitaxel

INTERVENTIONS:
Biological: bleomycin sulfate
Biological: filgrastim
Drug: cisplatin
Drug: etoposide
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known which regimen of combination chemotherapy may be more effective for germ cell cancer.

PURPOSE: This randomized phase II/III trial is studying two different regimens of combination chemotherapy and comparing how well they work in treating men with germ cell cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Phase II

* Compare the complete response rates in men with intermediate prognosis germ cell cancer treated with bleomycin, cisplatin, and etoposide (BEP) vs bleomycin, cisplatin, etoposide, and paclitaxel (T-BEP).
* Define the toxicity profile of T-BEP in these patients.

Phase III

* Compare the disease-free survival of patients treated with these regimens.
* Compare the complete response rates and overall survival of patients treated with these regimens.
* Compare symptoms and aspects of quality of life at baseline and after treatment in patients treated with these regimens.
* Compare the acute and intermediate (1-2 years) side effects of these regimens in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to histology (seminoma vs non-seminoma) and hospital. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive cisplatin IV and etoposide IV on days 1-5 and bleomycin IV on days 1, 8, and 15.
* Arm II: Patients receive cisplatin, etoposide, and bleomycin as in arm I and paclitaxel IV over 3 hours on day 1. Patients also receive filgrastim (G-CSF) subcutaneously on days 6-15.

In both arms, treatment repeats every 3 weeks for a total of 4 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed before treatment randomization and at 1 and 2 years after randomization.

Patients are followed monthly for 1 year, every 2 months for 1 year, every 3 months for 1 year, every 6 months for 1 year, and then annually thereafter.

PROJECTED ACCRUAL: A total of 84-164 patients (42-82 per treatment arm) will be accrued for the phase II study. A total of 498 patients (249 per treatment arm) will be accrued for the phase III study. Accrual will be completed within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven germ cell cancer

  * Seminoma
  * Non-seminoma
  * Combined
* Intermediate prognosis

  * Non-seminoma:

    * Testis/retroperitoneal primary
    * No non-pulmonary visceral metastases
    * Meets 1 of the following criteria:

      * Alpha-fetoprotein (AFP) 1,000- 10,000 IU/L
      * Human chorionic gonadotropin (hCG) 5,000-50,000 IU/L
      * Lactic dehydrogenase (LDH) 1.5 times-10 times upper limit of normal (ULN)
  * Seminoma:

    * Any primary site
    * Any LDH and HCG
    * AFP normal
    * Non-pulmonary visceral metastases present

PATIENT CHARACTERISTICS:

Age:

* 16 to 50

Sex:

* Male

Performance status:

* WHO 0-2

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.25 times ULN
* AST no greater than 2 times ULN

Renal:

* Creatinine clearance at least 40 mL/min (unless due to obstructive uropathy which can be relieved by nephrostomy)

Other:

* No pre-existing neuropathy
* No other malignancy except basal cell skin cancer
* No other serious illness or medical conditions incompatible with the protocol

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Ages: 16 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 498 (Estimated)
Dates: Start 1998-10

PRIMARY OUTCOMES:
Failure-free survival as measured by Logrank

SECONDARY OUTCOMES:
Response to treatment as measured by normalized markers without residual viable cancer after CT scan or surgery
Overall survival as measured by Logrank at end of each course, at 6 weeks after completion of study treatment, every 6 months up to year 5, and then annually thereafter
Disease-free survival as measured by Logrank at end of each course, at 6 weeks after completion of study treatment, every 6 months up to year 5, and then annually thereafter
Toxicity as measured by NCI-CTC v2.0 at end of each course, at 6 weeks after completion of study treatment, every 6 months up to year 5, and then annually thereafter
Quality of life as measured by Quality of Life Questionnaire Core 30 (QLQ-C30) at baseline, during treatment, and at years 1 and 2

CONTACTS AND LOCATIONS:
Overall Officials: Ronald De Wit, MD, PhD, Study Chair — Daniel Den Hoed Cancer Center at Erasmus Medical Center
Locations (69):
- Ludwig Boltzmann Institute for Applied Cancer Research at Kaiser Franz Josef Hospital, Vienna, Austria
- Belgium (3):
  - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - U.Z. Gasthuisberg, Leuven
- Denmark (2):
  - Aarhus Universitetshospital - Aarhus Sygehus, Aarhus
  - Rigshospitalet - Copenhagen University Hospital, Copenhagen
- France (3):
  - Centre Regional Francois Baclesse, Caen
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif
- Germany (20):
  - Charite - Universitaetsmedizin Berlin - Campus Benjamin Franklin, Berlin
  - Universitaetsklinikum Bonn, Bonn
  - St. Johannes Hospital - Medical Klinik II, Duisburg
  - Universitaetsklinikum Essen, Essen
  - Klinik Fuer Innere Medizin, Hematology/Oncology, Ernst Moritz Armdt Universitaet, Greifswald
  - Allgemeines Krankenhaus Hagen, Hagen
  - Universitaetsklinikum Halle, Halle
  - University Medical Center Hamburg - Eppendorf, Hamburg
  - Universitaetsklinikum des Saarlandes, Homburg
  - Klinikum Kassel, Kassel
  - Klinikum der Stadt Ludwigshafen am Rhein, Ludwigshafen am Rhein
  - Universitaetsklinkum Magdeburg der Otto-von-Guericke-Universitaet Magdeburg, Magdeburg
  - Klinikum der Stadt Mannheim, Mannheim
  - Universitaetsklinikum Giessen und Marburg GmbH - Marburg, Marburg
  - Klinikum Rechts Der Isar - Technische Universitaet Muenchen, Munich
  - Medizinische Klinik und Poliklinik A - Universitaetsklinikum Muenster, Münster
  - Klinikum Nuernberg - Klinikum Nord, Nuremberg
  - Klinikum der Universitaet Regensburg, Regensburg
  - Klinikum Schwerin, Schwerin
  - Southwest German Cancer Center at Eberhard-Karls-University, Tübingen
- National Institute of Oncology, Budapest, Hungary
- Assaf Harofeh Medical Center, Ẕerifin, Israel
- Ospedale di Circolo e Fondazione Macchi, Varese, Italy
- Netherlands (7):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Academisch Medisch Centrum at University of Amsterdam, Amsterdam
  - Leiden University Medical Center, Leiden
  - Universitair Medisch Centrum St. Radboud - Nijmegen, Nijmegen
  - University Medical Center Rotterdam at Erasmus Medical Center, Rotterdam
  - Daniel Den Hoed Cancer Center at Erasmus Medical Center, Rotterdam
  - University Medical Center Utrecht, Utrecht
- Norwegian Radium Hospital, Oslo, Norway
- Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology - Warsaw, Warsaw, Poland
- National Cancer Institute - Bratislava, Bratislava, Slovakia
- Spain (10):
  - Hospital de la Santa Cruz i Sant Pau, Barcelona
  - Vall d'Hebron University Hospital, Barcelona
  - Institut Catala D'Oncologia, Barcelona
  - Hospital Universitario San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Sant Joan de Reus, Reus
  - Hospital Universidad Virgen Del Rocio, Seville
  - Hospital Universitario La Fe, Valencia
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza
- United Kingdom (17):
  - Addenbrooke's Hospital, Cambridge, England
  - Gloucestershire Oncology Centre at Cheltenham General Hospital, Cheltenham, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Saint Bartholomew's Hospital, London, England
  - University College Hospital - London, London, England
  - Christie Hospital, Manchester, England
  - Nottingham City Hospital NHS Trust, Nottingham, England
  - Rosemere Cancer Centre at Royal Preston Hospital, Preston, England
  - Berkshire Cancer Centre at Royal Berkshire Hospital, Reading, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - Royal South Hants Hospital, Southampton, England
  - Royal Marsden - Surrey, Sutton, England
  - Southend University Hospital NHS Foundation Trust, Westcliff-on-Sea, England
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Western Infirmary, Glasgow, Scotland
  - Gartnavel General Hospital, Glasgow, Scotland
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales